## **Cover Page**

Official Title: Effect of Fan Therapy on Dyspnea Associated With Ticagrelor Administration

in Intensive Care Patients

**NCT Number:** Not yet assigned

Document Date: 18 July 2024

Prepared by: Emine Tuğba Yorulmaz, PhD Student

Supervised by: Asst. Prof. Arzu Erkoç

**Document Type**: Informed Consent Form

**Informed Consent Form** (ICF) – İngilizce

**Document Type**: Informed Consent Form (ICF)

**Document Date**: 18 July 2024

Subtitle: Voluntary Participation Form

# Informed Consent Form for Voluntary Participation in the Study

This research is being conducted by PhD student Emine Tuğba Yorulmaz from Istanbul University-Cerrahpaşa, Department of Medical Nursing, under the supervision of Asst. Prof. Arzu Erkoç, as part of her doctoral dissertation.

## **Purpose of the Study:**

To determine the effect of fan therapy in the management of ticagrelor-associated dyspnea.

#### **Procedures:**

Complete forms and use a handheld fan toward your face three times a day for 1–3 days as instructed.

Study lasts ~2 days. Study will terminate if severe shortness of breath occurs.

#### Confidentiality:

Participation is voluntary. No identifying info collected. Data analyzed collectively for research publications.

### Rights:

You can withdraw anytime without consequences. Inform study personnel if you choose to withdraw.

#### Contacts:

Faculty Member: Arzu Erkoç, Dept. Nursing, Email: arzu.erkoc@iuc.edu.tr

PhD student: Emine Tuğba Yorulmaz, Email: emine.yorulmaz@acibadem.edu.tr

#### **Consent Statement:**

| have read | the above a | and voluntarily | agree to | participate. |
|---------------|-------------|-----------------|----------|--------------|
| (Signature: ַ | | _ Date: | ) | |